CLINICAL TRIAL: NCT04588896
Title: Continuous Glucose Monitoring as an Adjunct to Lifestyle Modification in Individuals With Impaired Glucose Tolerance: a Randomised Controlled Trial
Brief Title: Continuous Glucose Monitoring as Adjunct to Lifestyle Modification in Prediabetes
Acronym: FlashLMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Elaine Chow, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FlashLMP
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2020-12

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGM+LMP (Experimental): Continuous glucose monitoring (CGM) for 8 weeks in conjunction with lifestyle modification
  Interventions: Device: Continuous glucose monitoring; Behavioral: Lifestyle modification programme
- LMP only (Other): Lifestyle modification only
  Interventions: Behavioral: Lifestyle modification programme

INTERVENTIONS:
Device: Continuous glucose monitoring — Abbott Freestyle Libre CGM for 8 weeks in adjunct to lifestyle modification programme
  Arms: CGM+LMP
Behavioral: Lifestyle modification programme — Lifestyle modification programme

SUMMARY:
This is a 12-month prospective, open-label, non-masked, two arm randomized controlled trial comparing intermittently-viewed continuous glucose monitoring (iCGM) in addition to lifestyle modification programme (LMP) as compared with a LMP alone in individulas with impaired glucose tolerance (IGT). Following informed consent, participants will undergo screening where a fasting glucose, 75g OGTT, HbA1c, fasting lipid profile along with comprehensive medical and drug history to confirm eligibility. At week 0, participants will be randomised to CGM plus LMP versus LMP alone. Both groups will receive individualized structured LMP programme delivered by a dietitian and a fitness instructor. Outcomes will be evaluated by laboratory tests, physical measurement, physical activity and dietary compliance and questionnaires at Month 0, 4, 8, 12.

ELIGIBILITY:
Inclusion Criteria:

1. Impaired glucose tolerance as defined by will be defined as per the American Diabetes Association criteria based on 75g oral glucose tolerance test (OGTT) 2-hour glucose of between 7.8 and less than 11 mmol/L
2. Male or female age ≥ 18 years old and ≤ 65 years old.
3. BMI 18 to 40kg/m2
4. Willingness, ability and commitment to comply with LMP
5. Able to use a CGM as judged by investigator
6. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a suitable study candidate.
7. Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

1. Currently pregnant, lactating, as demonstrated by a positive pregnancy test at screening or planning pregnancy
2. Known diabetes
3. Current or previous use of glucose-lowering or weight loss drugs
4. Concurrent participation in other weight loss or lifestyle intervention programmes
5. Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
6. Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
7. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
8. Extensive skin changes/diseases that preclude wearing the FGM on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
9. Known uncontrolled thyrotoxicosis
10. Current use of steroids
11. Have a known allergy to medical-grade adhesives
12. Known current or recent alcohol or drug abuse
13. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
14. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
1-hour glucose from OGTT | 12 months
  1-hour plasma glucose from a 75 g oral glucose tolerance test

SECONDARY OUTCOMES:
HbA1c | 12 months
  Between-group differences in HbA1c
Fasting plasma glucose | 12 months
  Between-group differences in fasting plasma glucose
Body weight | 12 months
  Between-group differences in body weight
Body mass index | 12 months
  Between-group differences in body mass index
Waist circumference | 12 months
  Between-group differences in waist circumference
3 day diet record | 12 months
  Differences in daily nutrient intake between groups
Physical activity levels | 12 months
  Daily number of steps as measured by a sealed pedometer
Socio-cognitive measures | 12 months
  Self-efficacy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No